CLINICAL TRIAL: NCT00003320
Title: Pilot Study of Adjuvant Fractionated Stereotactic Radiotherapy Following Surgical Removal of Cerebral Metastases
Brief Title: Radiation Therapy Following Surgery to Remove Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066270; UCLA-HSPC-970101503; UCLA-HSPC-970101502; NCI-G98-1416
Record Dates: First submitted 1999-11-01; First posted 2004-02-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: surgical procedure
Radiation: radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy after surgery to remove brain metastases may decrease the amount of radiation required to treat brain metastases.

PURPOSE: Pilot trial to study the effectiveness of radiation therapy following surgery to remove brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety and tolerability of focal stereotactic radiotherapy to the surgical bed following excision of cerebral metastases, as an alternative to whole brain irradiation. II. Measure the local relapse rate at the surgical site after surgery and stereotactic radiotherapy in patients with cerebral metastases. III. Measure the regional relapse rate, in the brain but away from the treated site, following treatment in these patients.

OUTLINE: All patients undergo surgical removal of their cerebral metastases followed by adjuvant fractionated stereotactic radiotherapy daily for 5 days. Patients are given up to 5 weeks following surgery to recover and reach the required performance status. Radiotherapy must commence within 6 weeks of surgery. Patients are followed at 2 weeks after treatment, monthly for 6 months, every 3 months for the next 18 months, every 6 months for the next year, and then annually for years 3-5.

PROJECTED ACCRUAL: There will be 20-40 patients accrued into this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cerebral metastases post surgical resection
* No greater than 3 cerebral metastases postresection
* Gross resection at operation as documented in operation note and postoperative MRI Patients must have current surgical sites that have not been previously irradiated
* No other indication for whole brain irradiation (i.e., multiple untreated metastases not suitable for single fraction stereotactic radiotherapy, leptomeningeal disease)
* Age: 18 and over
* Karnofsky 60-100%
* Life expectancy: At least 3 months
* Prior or concurrent required steroids allowed
* Prior stereotactic radiotherapy of cerebral metastases allowed provided no prior irradiation of current surgical sites
* Prior surgery of cerebral metastases allowed

Exclusion Criteria:

* severe asthma requiring therapy
* allergy to iodine or contrast media
* pregnant
* concurrent chemotherapy
* prior whole brain irradiation or focal irradiation to current sites of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1997-03; Primary Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Ford, MD, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States